CLINICAL TRIAL: NCT03894943
Title: Quantitative Sensory Testing and PET/CT Scanning in Assessment of Surgical Outcome for Lumbar Disc Herniation
Acronym: PET-Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spine Centre of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Christian Støttrup, PhD fellow, MD, Spine Centre of Southern Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: S-20140052
Record Dates: First submitted 2019-03-27; First posted 2019-03-29 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Lumbar Disc Herniation; Radiculopathy Lumbar
Keywords: PET/CT
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- General (Experimental): All subjects will undergo ordinary surgical treatment for their lumbar disc herniation. Experimentally, all subjects participating in the study will receive PET/CT scans and sensory testing as specified below.
  Interventions: Diagnostic Test: PET/CT scan; Diagnostic Test: Quantitative Sensory Testing

INTERVENTIONS:
Diagnostic Test: PET/CT scan — Patient receive a PET/CT scan of their cerebrum and lumbar spine prior to surgery, 4-6 weeks after surgery and 6 months after surgery
Diagnostic Test: Quantitative Sensory Testing — Patients undergo a battery of quantitative sensory tests prior to surgery, 4-6 weeks after surgery and 6 months after surgery

SUMMARY:
Patients with lumbar disc herniation suffer from pain and morbidity. Surgical intervention can be a quick and effective relief, however some individuals experience less favorable outcome.

This study tries to investigate and test the differences in pain perception and pain modulation between individuals. Using PET/CT scans the investigators try to visualize pain perception and -modulation in the CNS. This is subsequently correlated with a battery of pain tests and the surgical outcome of disc herniation surgery.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Clinical and radiological indication for LDH surgery, assessed by an experienced spinal surgeon
* Age 40-65 years
* Able to comply with regulations regarding medicine consumption (stated below)

Exclusion Criteria:

* History of previous spine surgery
* General contra-indication for spine surgery
* Greatly reduced kidney function
* Diagnosis of psychiatric disorder
* Current malignant disease
* History of radiation therapy
* Current chemotherapy
* History of spinal fracture
* Hematologic disease
* Current pregnancy or breast-feeding
* Chronic, generalized connective tissue disorders or chronic, non-specific pain disorders (fibromyalgia, whiplash (WAD I-V), etc.)

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
EuroQol-5D 3L | 1 year
  The 3-level version of EQ-5D (EQ-5D-3L) was introduced in 1990 by the EuroQol Group.
  The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement.
Oswestry Disability Index | 1 year
  The Oswestry Disability Index (also known as the Oswestry Low Back Pain Disability Questionnaire) is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools.
  0% to 20%: minimal disability: The patient can cope with most living activities.
  21%-40%: moderate disability: The patient experiences more pain and difficulty with sitting, lifting and standing. Travel and social life are more difficult, and they may be disabled from work. 41%-60%: severe disability: Pain remains the main problem in this group but activities of daily living is affected. These patients require a detailed investigation. 61%-80%: crippled: Back pain impinges on all aspects of the patient's life. 81%-100%: These patients are either bed-bound or exaggerating their symptoms.
Visual Analogue Scale | 1 year
  Both leg and back.
  Measure 0-100. 0 being no pain. 100 being worst imaginable pain.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Støttrup, MD, Principal Investigator — Sygehus Lillebælt

IPD SHARING:
Plan to Share IPD: Yes
Following completion of the study, data obtained during the research project will be made available to other researchers using Mendeleys sharing platform
Supporting Information: Study Protocol, Analytic Code
Time Frame: Will be shared late 2020

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-08): https://cdn.clinicaltrials.gov/large-docs/43/NCT03894943/Prot_SAP_000.pdf